CLINICAL TRIAL: NCT00076466
Title: Changes in Intracortical Inhibitory Processes Are Associated With the Development of Implicit Learning of a Motor Task
Brief Title: Brain Changes Associated With Learning a Motor Task
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040103; 04-N-0103
Record Dates: First submitted 2004-01-22; First posted 2004-01-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-14

CONDITIONS: Healthy
Keywords: Brain Excitability; Reaction Time; Plasticity; Motor Evoked Potential; Transcranial Magnetic Stimulation; Healthy Volunteer; HV

SUMMARY:
This study will determine: 1) whether learning a task with the dominant hand is accompanied by changes in the area of the brain that controls hand movement, and 2) how the brain is able to make these changes. Previous studies have shown that practicing a motor task can change brain excitability, but it is not known how well brain excitabilities are changed during motor learning. This study will measure changes in activity of the part of the brain that controls hand movement before, during, and after exercising the hand on a response pad.

Healthy normal volunteers between 18 and 40 years of age may be eligible for this study. Candidates who have not been evaluated at NIH within the past year will be screened with a brief interview about their current state of health and clinical and neurological examinations. Participants will undergo the following procedures:

Learning a finger movement/reaction time task

For this procedure, participants sit in front of a computer monitor with the index, middle, ring, and little fingers placed flat on four corresponding buttons of a response pad. They are asked to press one of the four buttons as fast as they can in response to an asterisk displayed on the monitor. The position of the asterisk indicates which button to push. Subjects perform nine sets of 120-button pushes with a 15-minute rest between each set. During the rest period, subjects undergo transcranial magnetic stimulation (described below), which causes twitches in the hand muscles. The electrical activity corresponding to the twitches is recorded by attaching electrodes (small metal disks) to the skin over the hand muscles.

Transcranial magnetic stimulation

For this test, an insulated wire coil is held over the scalp. A brief electrical current passes through the coil, creating a magnetic pulse that electrically stimulates the brain. The subject hears a click and may feel a pulling sensation on the scalp under the coil. The stimulation may also cause twitching in the muscles of the face, arm, or leg. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions.

...

DETAILED DESCRIPTION:
Objective: We aim to show that the development of implicit knowledge of a motor task is associated with decrease in intracortical GABA-related inhibition (ICI) in the trained muscles (accompanying increasing MEP amplitudes) and increase in ICI in non-trained neighboring muscles and that, after the knowledge becomes explicit, ICI modifications become less prominent.

It would be useful to know the role of ICI during learning. As some interventions or drugs are known to modify GABA activity, this study may even provide a rationale for using these interventions and drugs to enhance plastic changes in patients with impaired motor learning capabilities.

Several studies have shown that learning a motor task with one hand can be transferred to the contralateral hand (37, 43, 45, 46, 47). Studies have demonstrated that learning a finger sequence task (Serial Reaction Time test, SRTT) with the dominant-hand (trained) can be transferred to the contralateral hand (un-trained) (43,49,50). In this additional experiment we propose to investigate the effect of disrupting M1 (by using 1 Hz TMS, inhibitory effect) on motor learning in the trained hand (dominant) and in the un-trained hand (non-dominant). Evidence has shown that there is transcallosal connections between M1 of both hemispheres (40). Since M1 is active during implicit learning (41, 42) we expect 1 Hz TMS stimulation (inhibitory effect) over M1 will deteriorate implicit learning in the trained hand (dominant) as well as in the un-trained hand (non-dominant). This will be evaluated by assessing their effect on reaction times and accuracy of motor performance in both hands.

Study Population: 72 healthy volunteers, aged 18-40 will participate in the study. Subjects will be randomly assigned to either the test session or the control session.

Design: Subjects will complete a unique session. They will perform a serial-reaction-time task. The subjects will be instructed to push a button on a 4-button pad in response to a visual GO signal (which can appear at 4 different positions) using the appropriate digit and the appropriate button. There will be 9 blocks of 120 trials each. In the test group, in blocks 1, 4 and 7 the Go signal appears in a random order; in blocks 2-3, 5-6 and 8-9 the same 12-trial sequence is repeated 10 times. In the control group Go signals will appear in a random order in all blocks. Subjects won't be informed about the sequence but will be asked to notify anything they noticed about the task. If they do notice and report about a sequence they will be considered as having explicit knowledge. Between each block subjects will receive transcranial magnetic stimulations to assess ICI. ICI will be assessed on subjects at rest.

Outcome Measures: Behavioral effect of the motor training will be assessed by measuring the mean reaction times (RT) for digits II and V and the percentage of correct responses for each block.

Implicit learning will be assessed by the difference in RTs between block 3 and 4 and between block 6 and 7. Time at which explicit learning occurs will be assessed by verbal report and the degree of explicit learning by the number of correct items when repeating the sequence.

Implicit learning will be assessed in the trained hand (dominant) (see above) and in the un-trained hand. The un-trained hand will be tested by asking subjects to repeat two random blocks (familiarization) and two sequence blocks. One of these sequence blocks is a repetition of the same sequence that they learned with the dominant hand. The other sequence block is a new sequence containing the same number of characters as the previous sequence. Implicit learning on the un-trained hand will be assessed by the difference in RTs, between random block and the sequence block. In addition, implicit learning on the un-trained hand will be evaluated by testing the difference between the two sequence blocks repeated by the un-trained hand. The time at which explicit learning occurs will be assessed by verbal report and the degree of explicit learning by the number of correct items when repeating the sequence.

Intracortical inhibitory processes will be assessed by measuring the amount of ICI in trained muscles (first dorsal interosseus: FDI and adductor digit minimi: ADM) and a non-trained muscle (opponens pollicis brevis: OPB).

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal volunteers (aged 18 to 40 years) who are willing to participate and who have not participated yet in a protocol using a serial reaction time task (SRRT) and who are not or were not a piano player.

EXCLUSION CRITERIA:

Subjects with current use or history of alcohol or drug abuse, psychiatric disorder requiring hospitalization or prolonged treatment, head injury with loss of consciousness, epilepsy, and neurological disease. Subjects receiving drugs acting primarily on the central nervous system.

The following exclusion criteria are due to the use of trans cranial magnetic stimulation:

Subjects with cardiac pacemakers, intracardiac lines, implanted medication pumps.

Subjects with eye, blood vessel, cochlear, or eye implants, subjects with increased intracranial pressure as evaluated by clinical means, subjects with metal in the cranium except in the mouth, subjects with dental braces, metal fragments from occupational exposure or surgical clips in or near the brain.

Since this protocol utilizes paired pulse stimulation, there is no reason to exclude pregnant women. However, women in the last trimester of pregnancy will not be studied because they will likely be uncomfortable for three hours training.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72
Dates: Start 2004-01-22; Study Completion 2009-01-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bridgers SL, Delaney RC. Transcranial magnetic stimulation: an assessment of cognitive and other cerebral effects. Neurology. 1989 Mar;39(3):417-9. doi: 10.1212/wnl.39.3.417. PMID 2927652
- [Background] Butefisch CM, Davis BC, Wise SP, Sawaki L, Kopylev L, Classen J, Cohen LG. Mechanisms of use-dependent plasticity in the human motor cortex. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3661-5. doi: 10.1073/pnas.97.7.3661. PMID 10716702
- [Background] Classen J, Liepert J, Wise SP, Hallett M, Cohen LG. Rapid plasticity of human cortical movement representation induced by practice. J Neurophysiol. 1998 Feb;79(2):1117-23. doi: 10.1152/jn.1998.79.2.1117. PMID 9463469